CLINICAL TRIAL: NCT01493284
Title: Assessment Of The St. Jude Medical Portico™ Transcatheter Aortic Valve Implant (TAVI) And The SJM TAVI Transfemoral Delivery System (Portico TF EU)
Brief Title: Portico TAVI Implant With Transfemoral Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1105
Record Dates: First submitted 2011-12-05; First posted 2011-12-15 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: aortic stenosis; aortic valve stenosis; valvular heart disease; aortic valve replacement; transcatheter aortic valve implantation; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transfemoral Access (Experimental): Transfemoral Access for transcatheter aortic valve implant
  Interventions: Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Placement of the SJM Portico aortic valve with a transfemoral delivery system

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the SJM Portico Transcatheter Heart Valve and the SJM TAVI Transfemoral Transcatheter delivery system in subjects with severe symptomatic aortic stenosis (AS).

DETAILED DESCRIPTION:
Data will be collected at baseline, procedure, discharge, 30 days post implant, 3 months post implant, 6 months post implant, and 12 months post implant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written study Informed Consent for participation prior to procedure.
2. Subject is ≥ 18 years of age or legal age in host country.
3. Subject's aortic annulus diameter meets the range indicated in the Instructions for use as measured by echocardiogram (echo) or CT conducted within the past 90 days.
4. Subject has senile degenerative aortic stenosis with echocardiography (echo) derived mean gradient >40mmHg or jet velocity greater than 4.0 m/s or an initial valve area of <1.0 cm2 (or aortic valve area index ≤ 0.6 cm2/m2). (Baseline measurement taken by echo within 30 days of procedure).
5. Subject has symptomatic aortic stenosis as demonstrated by NYHA Functional Classification of II or greater.
6. Subject is deemed high operable risk and suitable for TAVI per the medical opinion of the Subject Selection Committee (See Section 3.1 for the definition of the Subject Selection Committee)
7. Subject's predicted operative mortality or serious, irreversible morbidity risk is <50% at 30 days.
8. In the opinion of the Subject Selection Committee and based upon angiographic measurements, the subject has suitable peripheral vessels and aorta to allow for access of the 18 French delivery system.
9. Subject has structurally normal cardiac anatomy.
10. Subject is willing and able to comply with all required follow-up evaluations.

Exclusion Criteria:

1. Subject has a history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months (≤180 days) of the index procedure.
2. Subject has carotid artery disease requiring intervention.
3. Subject has evidence of a myocardial infarction (MI) within the past 6 months (≤180 days) of the index procedure.
4. Subject has hypertrophic cardiomyopathy.
5. Subject has a native aortic valve that is congenitally unicuspid, bicuspid, quadricuspid or non-calcified as seen by echocardiography.
6. Subject has mitral or tricuspid valvular regurgitation (>grade III) or moderate to severe mitral stenosis.
7. Subject has aortic root angulation >70 degrees (horizontal aorta).
8. Subject has a pre-existing prosthetic valve or prosthetic ring in any position.
9. Subject refuses blood transfusion or surgical valve replacement.
10. Subject has left ventricular ejection fraction (LVEF) < 20%.
11. The subject has documented, untreated coronary artery disease (CAD) requiring revascularization.
12. Subject has severe basal septal hypertrophy.
13. Subject has had a percutaneous interventional or other invasive cardiac or peripheral procedure ≤ 14 days of the index procedure.
14. Subject has a history of or has active endocarditis.
15. Subject has echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
16. Subject has hemodynamic instability (requiring inotropic support or mechanical heart assistance).
17. Subject is in acute pulmonary edema or requiring intravenous diuretic therapy to stabilize heart failure.
18. Subject with significant pulmonary disease.
19. Subject has significant chronic steroid use.
20. Subject has a known hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
21. Subject has renal insufficiency as evidenced by a serum creatinine > 3.0 mg/dL (265µmol/L) or end-stage renal disease requiring chronic dialysis.
22. Subject has morbid obesity defined as BMI ≥ 40.
23. Subject's iliac arteries have severe calcification, tortuosity (>two 90 degree bends), diameter <6mm, or subject has had an aorto-femoral bypass.
24. Subject has ongoing infection or sepsis.
25. Subject has blood dyscrasias (leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy).
26. Subject has a current autoimmune disease that, in the opinion of the Principal Investigator precludes the subject from study participation.
27. Subject has significant aortic disease, including:

    * aortic abdominal aneurysm (AAA) ≥ 4cm
    * thoracic aneurysm (defined as a maximal luminal diameter of 5 cm or greater)
    * marked tortuosity
    * significant aortic arch atheroma or narrowing of the abdominal or thoracic aorta
    * severe tortuosity of the thoracic aorta.
28. Subject has a pre-existing endovascular stent graft in the supra- or infrarenal aorta or pre-existing stent grafts in the ileo-femoral arteries.
29. Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within the past 90 days prior to the index procedure.
30. Subject is currently participating in another investigational drug or device study.
31. Subject requires emergency surgery for any reason.
32. Subject has a life expectancy < 12 months.
33. Subject has other medical, social or psychological conditions that, in the opinion of the Subject Selection Committee, preclude the subject from study participation.
34. Subject is suffering from dementia or admitted to a chronic care facility which would fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits.
35. Subject has a known allergy to contrast media, nitinol alloys, porcine tissue, or bovine tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2011-12; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Manoharan, MD, Principal Investigator — Royal Victoria Hospital, Belfast
Locations (14):
- Adelaide Royal Hospital, Adelaide, Australia
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Germany (6):
  - Kerckhoff Klinik, Bad Nauheim
  - Heart Center Bernau, Bernau
  - Asklepios Klinik-St. Georg, Hamburg
  - Klinikum der Universität Jena, Jena
  - Klinik fur Herzhirurgie Karlruhe GmbH, Karlsruhe
  - Herzzentrum Leipzig, Leipzig
- Medical Center Leeuwarden, Leeuwarden, Netherlands
- United Kingdom (5):
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - Glenfield Hospital, Leicester
  - Kings College, London
  - St. Thomas' Hospital, London
  - Derriford Hospital, Plymouth, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walther T, Manoharan G, Linke A, Mollmann H, Holzhey D, Worthley SG, Kim WK, Schafer U. Incidence of new-onset left bundle branch block and predictors of new permanent pacemaker following transcatheter aortic valve replacement with the Portico valve. Eur J Cardiothorac Surg. 2018 Sep 1;54(3):467-474. doi: 10.1093/ejcts/ezy078. PMID 29534170
- [Derived] Linke A, Holzhey D, Mollmann H, Manoharan G, Schafer U, Frerker C, Worthley SG, van Boven AJ, Redwood S, Kovac J, Butter C, Sondergaard L, Lauten A, Schymik G, Walther T. Treatment of Aortic Stenosis With a Self-Expanding, Resheathable Transcatheter Valve: One-Year Results of the International Multicenter Portico Transcatheter Aortic Valve Implantation System Study. Circ Cardiovasc Interv. 2018 Feb;11(2):e005206. doi: 10.1161/CIRCINTERVENTIONS.117.005206. PMID 29444998

RESULTS

PARTICIPANT FLOW:
Groups:
- Transfemoral: Transfemoral access
Period: Overall Study
Arm/Group | Transfemoral
Started | 222
Completed | 161
Not Completed | 61
Not completed — Death | 29
Not completed — Withdrawal by Subject | 32

BASELINE CHARACTERISTICS:
Arm/Group | Transfemoral
Number analyzed (Participants) | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.0 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165
  Male | 57
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 15
  Denmark | 3
  United Kingdom | 48
  Australia | 15
  Germany | 141
STS risk score of mortality [Mean (Standard Deviation); unit: Percentage] — The Society of Thoracic Surgeons (STS) score measures patient risk of operative mortality and morbidity after adult cardiac surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  Percentage | 5.8 (3.3)
NYHA class III/IV [Count of Participants; unit: Participants] — NYHA Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  NYHA Class II: Subjects with cardiac disease resulting in slight limitation of physical activity.
  NYHA Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  NYHA Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Participants | 175
History of pulmonary hypertension [Count of Participants; unit: Participants] | 68
Porcelain aorta [Count of Participants; unit: Participants] | 8
History of atrial fibrillation [Count of Participants; unit: Participants] | 85
Renal failure/insufficiency [Count of Participants; unit: Participants] | 73

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Description: Number of participants that reported all cause mortality
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral
Number analyzed (Participants) | 222
Participants | 8

2. Secondary Outcome: Number of Select Cardiovascular Adverse Events
Description: Number of participants with select cardiovascular adverse events
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Transfemoral
Number analyzed (Participants) | 222
participants
  Cardiovascular death | 8
  Myocardial Infarction | 7
  Stage 3 Acute kidney injury | 3
  Disabling (major) stroke | 7
  Non-disabling (minor) stroke | 5
  Life threatening or disabling bleeding | 8

3. Secondary Outcome: Participant NYHA Classification at Day 30
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life.
  Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest.
  The Criteria Committee of the New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th ed. Boston, Mass: Little, Brown & Co; 1994:253-256.
Time Frame: day 30
Population: Analysis for participants that completed visit and assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral
Number analyzed (Participants) | 181
Participants
  NYHA 1 | 52
  NYHA II | 105
  NYHA III | 22
  NYHA IV | 2

4. Secondary Outcome: Number of Participants With Acute Device Success
Description: 1. Successful vascular access, delivery and deployment of the device and successful retrieval of the delivery system
  2. Correct position of the device in the proper anatomical location
  3. Intended performance of the prosthetic heart valve (Aortic Valve Area >1.2 cm2 and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, without moderate or severe prosthetic valve AR)
  4. Only one valve implanted in the proper anatomical location
Time Frame: 7 days
Population: Successful vascular access, delivery and deployment of the device
Measure: Count of Participants; unit: Participants
Arm/Group | Transfemoral
Number analyzed (Participants) | 222
Participants | 216

ADVERSE EVENTS:
Time Frame: 1-year
Arm/Group | Transfemoral
All-Cause Mortality (participants affected / at risk) | 29/222
Serious Adverse Events (participants affected / at risk) | 102/222
Other Adverse Events (participants affected / at risk) | 18/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transfemoral (N=222)
All-cause death (General disorders) | 29 (29)
Cardiovascular Death (Cardiac disorders) | 20 (20)
Myocardial infarction (Cardiac disorders) | 7 (7)
Stage 3 acute kidney injury (Renal and urinary disorders) | 6 (6)
Life-threatening or disabling bleeding (Vascular disorders) | 11 (11)
Disabling stroke (Renal and urinary disorders) | 12 (12)
Major vascular complications (Vascular disorders) | 19 (23)
Stage 1 acute kidney injury (Renal and urinary disorders) | 5 (5)
Stage 2 acute kidney injury (Renal and urinary disorders) | 2 (2)
Non-disabling stroke (Renal and urinary disorders) | 6 (6)
Pacemaker implantation (Cardiac disorders) | 33 (33)
Heart failure (Cardiac disorders) | 37 (47)
Coronary obstruction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transfemoral (N=222)
Hypertension (Cardiac disorders) | 7 (7)
Hyponatremia (Investigations) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes